CLINICAL TRIAL: NCT02425917
Title: Comparison of Intermittent Pneumatic Compression (IPC) of the Calf and gekoTM Neuromuscular Electrostimulation (NMES) Device on Lower Limb Circulation Following Elective Total Hip Replacement (THR)
Brief Title: IPC-CALF Versus GEKO in Post-op Total Hip Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not relevant to the sponsor
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FKD-IPC-002
Record Dates: First submitted 2015-04-14; First posted 2015-04-24 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-05

CONDITIONS: Total Hip Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- geko (Experimental)
  Interventions: Device: geko
- ipc-calf (Active Comparator): intermittent pneumatic compression of the calf
  Interventions: Device: IPC-Calf

INTERVENTIONS:
Device: geko — neuromuscular electrostimulator
  Arms: geko
Device: IPC-Calf — IPC used on calf with or without geko
  Arms: ipc-calf

SUMMARY:
This study is designed to compare the effect of IPC on post-operative circulation in lower limbs with gekoTM device after total hip replacement procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female
2. Aged over 18-80 years
3. Be in good general health and fitness other than the clinical requirement for a planned hip replacement.
4. Free of significant abnormal findings as determined by medical history (specifically an absence of DVT or haematological disorders.
5. No history or signs of drug abuse (including alcohol), licit or illicit.
6. Has not used any medications (prescribed or over-the-counter including herbal remedies) judged to be significant by the Principal Investigator (PI) during the thirty (30) days preceding the study.
7. Able to understand the Patient Information Sheet and willing to sign the written Informed Consent Form.
8. Able and willing to follow the protocol requirements.

Exclusion Criteria:

1. Are requiring hip revision surgery
2. History or signs of significant haematological disorders (especially in relation to clotting or coagulation or previous deep or superficial vein thrombosis/pulmonary embolism).
3. Significant Peripheral arterial disease (ABPI < 0.8), varicose veins or lower limb ulceration or ischemia.
4. Recent surgery within the last 3 months (such as abdominal, gynaecological, hip or knee replacement).
5. Recent trauma to lower limb.
6. Chronic Obesity (BMI Index >40kg/m2).
7. Pregnancy.
8. Significant history of following diseases i. Cardiovascular: Recent MI (< 6 months) ii. Percutaneous Coronary Intervention (PCI) with stent (< 3 months for Bare metal stent (BMS) and < 12 months for Drug Eluding Stent (DES) iii. Moderate to severe CCF, uncontrolled AF iv. Neurological: Stroke, Hemiplegia/Paraplegia, Myopathies v. Renal: Moderate to severely impaired renal function vi. Hepatic: Moderate to severely impaired hepatic function vii. Psychiatric disorders viii. Dermatological conditions affecting lower limbs ix. Haematological conditions i.e. coagulation disorders, sickle cell disease
9. A pulse rate of less than 40 beats/minute
10. A sitting systolic blood pressure >180 and <100 mmHg and/or a sitting diastolic pressure of >100 mmHg.
11. Any significant illness during the four (4) weeks preceding the hip replacement surgery.
12. Participation in any clinical study during the eight (8) weeks preceding the screening period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Ultra sound measurements of haemodynamics | 10mins

SECONDARY OUTCOMES:
Adverse event rate | 3 hrs
patient rated tolerability | 3 hrs
  A questionnaire has been designed to record the opinion of the patient with regard to both devices, in particular how comfortable the devices were to wear. The patient will be asked to rate how comfortable the devices are to wear on a scale of 1-5, 1 being very comfortable and 5 being extremely uncomfortable